CLINICAL TRIAL: NCT05142514
Title: A Phase IIb Study to Evaluate Safety and Immunogenicity of Recombinant Protein RBD Fusion Dimer Candidate Vaccine Against the Virus That Cause COVID-19, Known as Severe Acute Respiratoy Syndrome Coronavirus 2 (SARS-CoV-2) in Adult Healthy Volunteers
Brief Title: Safety and Immunogenicity of Recombinant Protein RBD Fusion Dimer Vaccine Against the Virus That Cause COVID-19, Known as Severe Acute Respiratoy Syndrome Coronavirus 2 (SARS-CoV-2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hipra Scientific, S.L.U (Industry)
Collaborators: Laboratorios Hipra, S.A. (Industry); National Institute of Hygiene and Epidemiology, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: HAN-01
Record Dates: First submitted 2021-11-17; First posted 2021-12-02 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; SARS-CoV-2 Acute Respiratory Disease
MeSH Terms: conditions — COVID-19 | interventions — HIPRA COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 Vaccine HIPRA (Experimental): Subjects will receive 2 injections of COVID-19 vaccine HIPRA administered 21 days apart.
  Interventions: Biological: COVID-19 Vaccine HIPRA
- Commercial COVID-19 Vaccine (Active Comparator): Subjects will receive 2 injections of COVID-19 vaccine HIPRA administered 21 days apart
  Interventions: Biological: Cominarty (Pfizer-BioNtech)

INTERVENTIONS:
Biological: COVID-19 Vaccine HIPRA — Subjects will receive 2 injections of COVID-19 vaccine HIPRA administered 21 days apart
  Arms: COVID-19 Vaccine HIPRA
Biological: Cominarty (Pfizer-BioNtech) — Subjects will receive 2 injections of Cominarty administered 21 days apart
  Arms: Commercial COVID-19 Vaccine

SUMMARY:
This is a Phase IIb, randomized, controlled, observer-blinded, clinical trial to evaluate safety and immunogenicity of COVID-19 Vaccine HIPRA in adult healthy volunteers in Vietnam

DETAILED DESCRIPTION:
The study population includes 256 healthy adults aged 18-60 which will be randomized in a ratio 1:1 test:commercial vaccine. Each participant will receive 2 immunisations separated by 21 days and will be followed for 24 weeks after the second dose.

ELIGIBILITY:
Inclusion Criteria:

* Adults males or females between 18-60 years of age at the day of screening.
* Willing and able to comply with scheduled visits, laboratory test, complete diaries and other study procedures.
* Body Mass Index 18 to 40 Kg/m2 at screening.
* COVID19 negative quick test or PCR test and negative serum IgG binding antibody response to the SARS-CoV-2 S glycoprotein at screening or prior the first vaccination. If an enrolled subject has neutralizing antibodies at baseline, he or she will be excluded from final analysis.
* Willing to avoid all other vaccines within 4 weeks before and after each injection. Seasonal influenza vaccination is allowed if it is received at least 14 days before or after the vaccination.
* Women of childbearing potential must have a negative pregnancy test in urine before the inclusion of the study and prior to each vaccination.
* If female of childbearing potential, willing to use highly effective contraceptive methods or have practiced sexual abstinence from the screening visit until 8 weeks after the last injection.
* If male and not sterilized, willing to avoid impregnating female partners from screening until 8 weeks after last injection.
* Willing and able to provide written informed consent prior the initiation of any study procedures.

Exclusion Criteria:

* Pregnant or lactating or intending to become pregnant or plans to breastfeed during the study.
* Positive pregnancy test at screening or prior to each vaccination.
* Any medical disease (acute, subacute, intermittent or chronic) or condition with grade 2 or above that in the opinion of the investigator compromise the volunteer's safety, preclude vaccination or compromise interpretation of the results.
* History of serious psychiatric condition likely to affect participation in the study.
* History of respiratory disease (e.g., chronic obstructive pulmonary disease (COPD) and asthma) requiring any daily medications currently or any treatment of respiratory disease exacerbations (e.g., asthma exacerbation) in the last 5 years.
* History of significant cardiovascular disease including hypertension (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease) or history of myocarditis or pericarditis as an adult.
* History of neurological or neurodevelopmental conditions (e.g., migraines, epilepsy, stroke, seizures in the last 3 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis or transverse myelitis).
* Ongoing malignancy or recent diagnosis of malignancy in the last five years excluding basal cell and squamous cell carcinoma of the skin, which are allowed.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent severe infections.
* Any autoimmune or immunodeficiency disease/condition (iatrogenic or congenital).
* Acute illness within 72 hours prior each vaccination that in the opinion of the investigator may interfere the evaluation of safety parameters.
* Usage of any investigational drug ≤ 90 days prior to study entry or plan to participate in another research involving an investigational product (drug/biologic/device) within 12 months after the first study vaccination.
* History of hypersensitivity or severe allergic reaction including anaphylaxis, generalized urticarial, angioedema and other significant reactions related to food, drugs, vaccines or pharmaceutical agents.
* History of allergic disease or reactions likely to be exacerbated by any component of the COVID-19 vaccine HIPRA
* Use of any immunosuppressant, glucocorticoids, or other immune-modifying drugs within 2 months prior to first study vaccination; or anticipation of the need for immunosuppressive treatment within 6 months after last vaccination.
* Received immunoglobulin, blood-derived products, or other immunosuppressant drugs within 90 days prior to first study vaccination.
* Known disturbance of coagulation (iatrogenic or congenital) or blood dyscrasias.
* Known bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture.
* Chronic liver disease
* Positive test for HIV types 1 or 2 infection, hepatitis B surface antigen (HBsAg), or hepatitis C virus antibodies (HCV Abs) at screening
* Suspected or known current alcohol abuse or any other substances abuse (except tobacco).
* History of COVID-19 infection.
* Receipt of medications intended to prevent COVID-19.
* Ever received an experimental vaccine against COVID-19.
* Close contact of anyone known to have SARS-CoV-2 infection within 15 days prior to screening visit.
* Being directly involved in the conduct of the study
* Any condition and/or laboratory finding that at the investigator consideration would interfere with the study or put at risk the participant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 629 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of COVID-19 HIPRA vaccine in healthy adult volunteers | 7 days
  Number and percentage of solicited local and systemic reactogenicity adverse events for 7 days following each vaccination.
Safety and tolerability of COVID-19 HIPRA vaccine in healthy adult volunteers | 28 days
  Number and percentage of unsolicited local and systemic reactogenicity adverse events for 28 days following each vaccination.
Safety and tolerability of COVID-19 HIPRA vaccine in healthy adult volunteers | 7 days
  Change from baseline in safety laboratory parameters at 7 days following each vaccination.
Safety and tolerability of COVID-19 HIPRA vaccine in healthy adult volunteers | 30 weeks
  Number and percentage of serious adverse events throughout the study duration.
Safety and tolerability of COVID-19 HIPRA vaccine in healthy adult volunteers | 30 weeks
  Number and percentage of adverse events of special interest (AESI) throughout the study duration.
Safety and tolerability of COVID-19 HIPRA vaccine in healthy adult volunteers | 30 weeks
  Number and percentage of medically attended adverse events (MAAE) related to study vaccine throughout the study duration.

SECONDARY OUTCOMES:
Immunogenicity | Day 21 and 35.
  Neutralization titer for each individual sample and GMT for group comparison at Day 21 and 35.
Immunogenicity | Day 21 and 35.
  IC50 of beta and delta variants.
Immunogenicity | Day 21 and 35.
  Geometric mean fold rise (GMFR) in neutralizing antibodies titers from baseline at Day 21 and 35.
Immunogenicity at long-term | 24 and 48 weeks after the second dose
  Neutralization titer for each individual sample and GMT for group comparison at 24 and 48 weeks after the second dose.
Immunogenicity at long-term | 24 weeks after the second dose
  IC50 of beta and delta variants.
Immunogenicity at long-term | 24 weeks after the second dose
  GMFR in neutralizing antibodies titers from baseline at 24 weeks after the second dose.
Immunogenicity to the SARS-CoV-2 spike glycoprotein | Day 21 and 35
  Total binding antibody titer and GMT for group comparison at Day 21 and 35.
Immunogenicity to the SARS-CoV-2 spike glycoprotein | Day 21 and 35
  GMFR in total binding antibodies titer from baseline at Day 21 and 35.
Immunogenicity to the SARS-CoV-2 spike glycoprotein at long-term | 24 weeks after the second dose
  Total Binding antibody titer and GMT for group comparison at 24 weeks after the second dose.
Immunogenicity to the SARS-CoV-2 spike glycoprotein at long-term | 24 weeks after the second dose
  GMFR in total binding antibodies titer from baseline at 24 weeks after the second dose.
Immunogenicity to the SARS-CoV-2 spike glycoprotein | Day 21 and 35.
  Percentage of subjects who seroconverted defined as a ≥4-fold change in total binding antibody titer from baseline at Day 21 and 35.

OTHER OUTCOMES:
Number of participants with symptomatic SARS-CoV-2 infections in participants without evidence of infection before COVID-19 HIPRA vaccination. | 30 weeks
  Number and percentage of subjects with symptomatic SARS-CoV-2 infections according to COVID-19 infection criteria.
Number of COVID-19 severe infections after receiving COVID-19 HIPRA vaccine. | 30 weeks
  Number and percentage of COVID-19 severe infections throughout the study duration.
Number of COVID-19 severe infections after receiving COVID-19 HIPRA vaccine. | 30 weeks
  Number and percentage of hospital admissions associated with COVID-19 throughout the study duration.
Number of COVID-19 severe infections after receiving COVID-19 HIPRA vaccine. | 30 weeks
  Number and percentage of intensive care unit (ICU) admissions associated with COVID-19 throughout the study duration.
Number of COVID-19 severe infections after receiving COVID-19 HIPRA vaccine. | 30 weeks
  Number and percentage of deaths associated with COVID-19 throughout the study duration.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Hygiene and Epidemiology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No